CLINICAL TRIAL: NCT01459211
Title: A Pilot Study to Establish the Safety & Efficacy of a Combination of Dexamethasone & Lenalidomide in Patients With Relapsed/Refractory Chronic Lymphocytic Leukaemia (CLL)
Brief Title: Pilot Study to Establish Safety & Efficacy of a Combination of Dexamethasone and Lenalidomide in Patients With Relapsed or Refractory Chronic Lymphocytic Leukaemia (CLL)
Acronym: LenD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/09/387
Record Dates: First submitted 2011-10-18; First posted 2011-10-25 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide & Dexamethasone (Other): Lenalidomide, 5mg daily, increased to 10mg after 1st cycle. Dexamethasone, 20mg days 1-4 each cycle
  Interventions: Drug: Lenalidomide & Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide & Dexamethasone — Subjects with relapsed or refractory CLL will receive twelve 28-day cycles of treatment. Each cycle will consist of:
  1. Oral Dexamethasone (20mg daily, days 1-4),
  2. Oral Lenalidomide on days 1-28 of each cycle, starting at 5mg per day in cycle 1 in patients with creatinine clearance ≥ 60ml/min calculated by Cockcroft-Gault. The dose will be increased to 10mg per day with cycles 2-12 unless there is evidence of disease progression or unacceptable drug toxicity
  Other Names: Revlimid

SUMMARY:
The purpose of this study is to establish the safety and efficacy of a combination of dexamethasone and lenalidomide (Revlimid®) (D+L) in subjects with relapsed or refractory CLL who have failed or are unable to tolerate standard up-front therapy with regimens containing Fludarabine or in those with mutations in the p53 gene, CAMPATH-1H.

DETAILED DESCRIPTION:
In this study we plan to assess the safety and tolerability of the combination of dexamethasone, and lenalidomide (D+L) in patients with relapsed or refractory CLL, a subgroup with limited treatment options. Lenalidomide offers an alternative way of treating CLL. In a Phase 1 safety and pharmacokinetics study (study 1398/180) in healthy male volunteers, it was demonstrated that lenalidomide administered at a dose of 100 mg twice a day for 6 days had an acceptable safety profile with grade 1-2 rash and pruritus being the primary adverse events associated with the administration of the compound. In myeloma and MDS, lenalidomide has been studied mostly at two doses: 25 mg/day and 10 mg/day. In CLL significant toxicity was observed with these two dose levels, including tumour lysis syndrome and tumour flare.47,48 We therefore plan to start therapy with lenalidomide at a relatively low dose of 5mg/day, days 1-28, with cycle 1 and escalate to the maximum dose of 10mg/day with cycles 2-12. We have elected to administer lenalidomide continuously as opposed to pulsing over 14-21 days of each cycle to reduce the risk of tumour flare reaction (TFR), when this agent is reintroduced with each cycle. Finally, lenalidomide will be administered in combination with Dexamethasone, at a dose of 20mg/day for 4 days in each 28 day cycle as this allows convenient oral administration. We and others have demonstrated that Dexamethasone level is effective in CLL patients who are refractory or have relapsed following primary Fludarabine therapy. The combination of D+L will likely reduce toxicity, especially TFR, whilst improving overall efficacy without promoting the emergence of chemoresistant clones in which tumour suppressor genes have been inactivated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed or refractory CLL as defined by the NCIWG criteria, requiring treatment
* 1-3 lines of prior therapy
* Fludarabine- or Alemtuzumab-based therapy inappropriate
* WHO Performance status ≤2
* Age ≥ 18 years
* Life expectancy > 6 months
* Male and female subjects must meet the inclusion criteria for the Lenalidomide Pregnancy Prevention Risk Management Plan.
* Male and female subjects must agree to follow the Lenalidomide Pregnancy Prevention Risk Management Plan (including contraception 4 weeks before, during and 4 weeks after treatment for females of child-bearing potential).
* Signed informed consent

Exclusion Criteria:

* Previously untreated CLL
* Fit patients for whom alemtuzumab or fludarabine- based therapy would be appropriate
* Creatinine clearance < 30ml/min calculated by Cockcroft-Gault
* Bilirubin > 1.5 x upper limit of normal
* Patients with marrow suppression resulting in significant cytopenia (Neutrophils <0.5 x 109/l, Platelets <30 x 109/l).
* Radiotherapy, radioimmunotherapy, biological therapy, chemotherapy or other investigational therapy within 4 weeks prior to study Day 1.
* Known infection with HIV, hepatitis B or hepatitis C.
* Uncontrolled glaucoma, diabetes mellitus, hypertension or symptomatic peptic ulcer disease
* Peripheral neuropathy > grade 1
* Proven or suspected transformation to aggressive B-cell malignancy (e.g. large -B-cell lymphoma, Richter's syndrome, or PLL).
* Second malignancy requiring treatment other than non metastatic skin or prostate tumours
* Any medical condition that would require long-term use (>1 month) of systemic corticosteroids at a dose greater than 5mg/day of prednisolone during study treatment.
* Active uncontrolled bacterial, viral or fungal infections Cardiac failure, myocardial infarction within 6 months prior to study day 1, or evidence of ischaemia on ECG within 30 days prior to study day 1.
* Epileptic disorders requiring anticonvulsant therapy
* Major surgery, other than diagnostic surgery within 4 weeks prior to Study Day 1.
* Pregnant or currently breastfeeding.
* Patients who for other reasons are not expected to complete the study
* Subjects with a known allergy to allopurinol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who achieve objective response (CR + PR) according to the updated 1996 NCIWG criteria measured at 4 weeks after the completion of chemotherapy | 4 weeks after the completion of chemotherapy

SECONDARY OUTCOMES:
Duration of response | Time from initial response to first relapse/progression or death
  Response will be assessed 4 weeks after completion or discontinuation of treatment. Response and disease status will be assessed at monthly follow up visits until 6 months post completion or discontinuation of treatment. After this patients will be assessed annually until death and the date of first relapse or progression will be recorded for every patient, therefore giving a duration of response in months.
Time to next treatment | Time from end of chemotherapy to next treatment
  Patients will be assessed after completion or discontinuation of treatment monthly until 6 months, and then assessed annually. At these assessments the patients status will be assessed and any further treatment for the disease will be recorded and the date of this treatment. Therefore the time from end of chemotherapy to next treatment will be recorded for each patient, in months.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Nathwani, Principal Investigator — University College, London
Locations (2):
- United Kingdom (2):
  - Royal Liverpool University Hospital, Liverpool
  - University College London, London

IPD SHARING:
Plan to Share IPD: Undecided